CLINICAL TRIAL: NCT04003402
Title: A Phase 1 Randomized, Placebo-controlled, Crossover Study to Assess Potential Interaction Between ASP8062 and Alcohol in Healthy Adult Subjects
Brief Title: A Study to Assess Potential Interaction Between ASP8062 and Alcohol in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 8062-CL-2001
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: alcohol effect; Healthy Volunteer; ASP8062
MeSH Terms: interventions — ASP8062; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1: Participants receiving treatment sequence A,B,C,D (Experimental): Eligible participants will received treatment sequence A, B, C, D. Each participant will receive a single oral dose and each treatment period has a minimum of a 14 day washout period between investigational product administration.
  A= ASP8062 with Alcohol; B= ASP8062 with Placebo Alcohol; C= Placebo ASP8062 with Alcohol; D = Placebo ASP8062 with Placebo Alcohol
  Interventions: Drug: ASP8062; Drug: Alcohol; Drug: ASP8062 Placebo; Drug: Alcohol Placebo
- Sequence 2: Participants receiving treatment sequence B,D,A,C (Experimental): Eligible participants will received treatment sequence B, D, A, C. Each participant will receive a single oral dose and each treatment period has a minimum of a 14 day washout period between investigational product administration.
  B= ASP8062 with Placebo Alcohol; D = Placebo ASP8062 with Placebo Alcohol; A= ASP8062 with Alcohol; C= Placebo ASP8062 with Alcohol
  Interventions: Drug: ASP8062; Drug: Alcohol; Drug: ASP8062 Placebo; Drug: Alcohol Placebo
- Sequence 3: Participants receiving treatment sequence C,A,D,B (Experimental): Eligible participants will received treatment sequence C, A, D, B. Each participant will receive a single oral dose and each treatment period has a minimum of a 14 day washout period between investigational product administration.
  C= Placebo ASP8062 with Alcohol; A= ASP8062 with Alcohol; D = Placebo ASP8062 with Placebo Alcohol; B= ASP8062 with Placebo Alcohol
  Interventions: Drug: ASP8062; Drug: Alcohol; Drug: ASP8062 Placebo; Drug: Alcohol Placebo
- Sequence 4: Participants receiving treatment sequence D,C,B,A (Experimental): Eligible participants will received treatment sequence D, C, B, A. Each participant will receive a single oral dose and each treatment period has a minimum of a 14 day washout period between investigational product administration.
  D = Placebo ASP8062 with Placebo Alcohol; C= Placebo ASP8062 with Alcohol; B= ASP8062 with Placebo Alcohol; A= ASP8062 with Alcohol
  Interventions: Drug: ASP8062; Drug: Alcohol; Drug: ASP8062 Placebo; Drug: Alcohol Placebo

INTERVENTIONS:
Drug: ASP8062 — oral
Drug: Alcohol — oral
  Other Names: ethanol
Drug: ASP8062 Placebo — oral
Drug: Alcohol Placebo — oral

SUMMARY:
The purpose of this study is to assess the potential for pharmacokinetic (PK) and pharmacodynamics (PD) interactions between ASP8062 and alcohol.

This study will also assess safety and tolerability of a single dose of ASP8062 with or without alcohol.

DETAILED DESCRIPTION:
Participants will be admitted to the clinical unit on day -1 of each period and will be residential for 6 days/5 nights. Participants will be discharged from the clinical unit on day 5 of each period on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit. Participants will return to the clinical unit on days 7 and 10 for pharmacokinetic blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female subjects (21 to 55 years of age, inclusive) who currently consume alcohol regularly but do not meet the diagnostic and statistical manual of mental disorders (DSM-5) criteria for alcohol use disorders and are able to consume 3 to 4 standard drinks at 1 occasion without causing excessive intoxication.
* Subject currently consumes alcohol regularly but does not meet the diagnostic and statistical manual of mental disorders (DSM-5) criteria for alcohol use disorders and subject is able to consume 3 to 4 standard drinks at 1 occasion without causing excessive intoxication. (note: standard drink =1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor).
* Subject has a body mass index (BMI) range of 18.5 to 32.0 kg/m2, inclusive and weighs at least 50 kg at screening.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 28 days after final investigational product (IP) administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 28 days after final IP administration.
* Female subject must not donate ova starting at first dose of IP and throughout the study period and for 28 days after final IP administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception, throughout the treatment period and for 90 days after final IP administration.
* Male subject must not donate sperm during the treatment period and for 90 days after final IP administration.
* Male subject with a pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 90 days after final IP administration.
* Subject agrees to not participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP8062, alcohol or any components of the formulations used.
* Subject has had previous exposure with ASP8062.
* Subject has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase and total bilirubin [TBL]) above 1.5 × upper limit of normal (ULN) on day -1 of period 1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has a current, untreated moderate or severe mental illness as assessed by the Mini International Neuropsychiatric Interview (MINI).
* Subject has a relevant history of suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 12 months or subject who is at significant risk to commit suicide using the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening and on day -1 of period 1.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Subject has a mean QT interval using Fridericia's correction formula (QTcF) of > 430 msec (for male subjects) and > 450 msec (for female subjects) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first IP administration, except for occasional use of paracetamol (up to 2 g/day), topical dermatological products, including corticosteroid products, hormonal contraceptives and hormone replacement therapy (HRT).
* Subject has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening or the subject tests positive for cotinine at screening.
* Subject has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening or the subject tests positive for alcohol at screening or on day -1 of period 1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the subject tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1 of period 1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B core antibodies, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ASP8062 in plasma: area under the concentration time curve from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 10 of each treatment period
  AUCinf will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ASP8062 in plasma: maximum concentration (Cmax) | Up to Day 10 of each treatment period
  Cmax will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of alcohol in Ethanol plasma: AUClast | Day 1 of each treatment period
  AUClast will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of alcohol in Ethanol plasma: Cmax | Day 1 of each treatment period
  Cmax will be recorded from the pharmacokinetic (PK) plasma samples collected.
Change from baseline in reaction times defined by Cogstate battery: psychomotor function | Baseline and Day 1 of each treatment period (90 minutes, 2.5 hours, 4 hours and 6 hours post dose)
  The psychomotor function domain will be assessed using the Detection Test. Participants will tap a moving target on a grid and reaction times will be recorded. Change from baseline will be reported at indicated time points. Lower scores mean better performance.
Change from baseline in reaction times defined by Cogstate battery: attention | Baseline and Day 1 of each treatment period (90 minutes, 2.5 hours, 4 hours and 6 hours post dose)
  The attention domain will be assessed using the Identification Test. Participants will answer "yes" or "no" to the question "is the card red or not?" and reaction times will be recorded. Change from baseline will be reported at indicated time points. Lower scores mean better performance.
Change from baseline in reaction times defined by Cogstate battery: working memory | Baseline and Day 1 of each treatment period (90 minutes, 2.5 hours, 4 hours and 6 hours post dose)
  The working memory domain will be assessed using the One Back Test. Participants will answer "yes" or "no" to the question "is the previous card the same?" and reaction times will be recorded. Change from baseline will be reported at indicated time points. Lower scores mean better performance.
Change from baseline in number of error attempts defined by Cogstate battery: executive function | Baseline and Day 1 of each treatment period (90 minutes, 2.5 hours, 4 hours and 6 hours post dose)
  The executive function domain will be assessed using the Groton Maze Learning Test. Participants will be asked to find a hidden pathway and the total number of errors made while attempting to learn the same pathway will be recorded. Change from baseline will be reported at indicated time points. Lower scores mean better performance.
Postural stability test assessed via the single-leg stance test | Day 1 of each treatment period
  Limb dominance will be determined and recorded prior to performing the single leg stance test. Time will commence when eyes are closed and end for any of the following reasons: participant uses arms; participant uses the raised foot; participant moves the weight bearing foot to maintain balance; a maximum of 45 seconds has elapsed; or participant opens eyes. The test will be repeated 3 times and each time will be recorded. The best and the average of the 3 trials will also be recorded.

SECONDARY OUTCOMES:
Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to 55 Days (End of Study)
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered an Investigational Product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 55 Days (End of Study)
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to 55 Days (End of Study)
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to 55 Days (End of Study)
  Number of participants with potentially clinically significant ECG values.
Number of participants with suicidal ideation and/or behavior as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Day 1 of each treatment period
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) will be reported.
Number of participants with Blood oxygen saturation (SpO2) level abnormalities and/or Adverse Events (AEs) | Day 1 of each treatment period
  Number of participants with potentially clinically significant SpO2 values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel International - EPCU Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.